CLINICAL TRIAL: NCT04931134
Title: Trigeminal Nerve Stimulation in Anxiety Disorders: a Randomized Controlled Trial
Brief Title: Treatment of Anxiety Disorders With Trigeminal Nerve Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Rafael Freire (Other)
Responsible Party: Sponsor-Investigator, Dr. Rafael Freire, Associate Professor, Department of Psychiatry, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6028648
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Panic Disorder; Generalized Anxiety Disorder; Social Anxiety Disorder
MeSH Terms: conditions — Panic Disorder; Generalized Anxiety Disorder; Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sham stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active stimulation (Experimental): Active or sham TNS treatment will be performed at the patients' home for approximately 8 hours per night 7 days a week for 8 consecutive weeks.
  Trigeminal nerve stimulation will occur by placement of electrodes (1.25" silver electrodes Bio-Flex BF4, Biotens/Vermed, Buffalo, NY, USA) bilaterally on the V1 branches of the trigeminal nerve (CNV) located on the forehead. Current will be generated from the EMS 7500 stimulator (TENS Products, Inc., Granby, CO) (Class II medical device) and will be set to a level that is clearly perceptible by each patient (i.e. tingling sensation) but not uncomfortable or painful. Current level will be determined for each patient at baseline and will likely be between 4-6 mA. Active stimulation will occur at 120 Hz with a 250 µs pulse width and with a duty cycle of 30 seconds on to 30 seconds off.
  Interventions: Device: Trigeminal nerve stimulation - active
- Sham stimulation (Sham Comparator): Active or sham TNS treatment will be performed at the patients' home for approximately 8 hours per night 7 days a week for 8 consecutive weeks.
  Sham stimulation will occur by placement of electrodes (1.25" silver electrodes Bio-Flex BF4, Biotens/Vermed, Buffalo, NY, USA) bilaterally on the V1 branches of the trigeminal nerve (CNV) located on the forehead. Current will be generated from the EMS 7500 stimulator (TENS Products, Inc., Granby, CO) (Class II medical device) and will be set to a level that is clearly perceptible by each patient (i.e. tingling sensation) but not uncomfortable or painful. Current level will be determined for each patient at baseline and will likely be between 4-6 mA. Sham stimulation will use the same parameters of active stimulation, but after 60 seconds the stimulator will turn off.
  Interventions: Device: Trigeminal nerve stimulation - sham

INTERVENTIONS:
Device: Trigeminal nerve stimulation - active — Active trigeminal nerve stimulation
  Arms: Active stimulation
Device: Trigeminal nerve stimulation - sham — Sham trigeminal nerve stimulation
  Arms: Sham stimulation

SUMMARY:
Primary objectives: The primary objective is to ascertain if trigeminal nerve stimulation is an effective treatment with high tolerability for patients with panic disorder, generalized anxiety disorder and social anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM5 criteria for panic disorder, social anxiety disorder or generalized anxiety disorder.

Exclusion Criteria:

* Subjects undergoing cognitive behavioural therapy.
* Subjects undergoing pharmacological treatment for an anxiety disorder.
* Subjects undergoing pharmacological treatment with antidepressants or benzodiazepines.
* Subjects with moderate to severe major depressive disorder based on the PHQ-9 test (score of 15 or above) at baseline.
* Moderate to high current suicidality or "suicide likely in near future" or current suicidal behavior disorder.
* Concurrent diagnosis of OCD, PTSD, bipolar disorder, schizophrenia, schizoaffective disorder, personality disorders, substance use disorders, intellectual disabilities or dementia.
* Subjects diagnosed with neurological diseases including trigeminal neuralgia.
* Pregnant or breastfeeding women.
* Subjects who are experiencing seizures.
* Individuals with implanted VNS or other electrical devices.
* Subjects who are already undergoing transcutaneous electrical nerve stimulation.
* Consumption of cannabis, any cannabis by-products, illicit drugs, or alcohol above 3 drinks per week.
* Consumption of natural health products that may affect anxiety or depression symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Response | Clinical Global Impression - Improvement scale (CGI-I) will be administered after 8 weeks of treatment.
  Treatment response will be defined as a score of 1 or 2 on the Clinical Global Impression - Improvement scale (CGI-I). CGI-I scores range from 0 to 7. Zero corresponds to "not assessed". Low scores correspond to improvement, high scores correspond to worsening.
Remission | Clinical Global Impression - Severity scale (CGI-S) will be administered after 8 weeks of treatment.
  Remission will be defined as a score of 1 or 2 on the Clinical Global Impression - Severity scale (CGI-S). CGI-S scores range from 0 to 7. Zero corresponds to "not assessed". Low scores correspond to mild and high scores correspond to severe.

SECONDARY OUTCOMES:
Generalized anxiety disorder symptoms | Generalized Anxiety Disorder 7-item scale (GAD-7) will be administered after 8 weeks of treatment.
  Improvement of generalized anxiety disorder symptoms measured with the Generalized Anxiety Disorder 7-item scale (GAD-7). Scores go from 0 (no generalized anxiety symptoms) to 21 (severe generalized anxiety symptoms).
Social anxiety disorder symptoms | Social Phobia Inventory (SPIN) will be administered after 8 weeks of treatment.
  Improvement of social anxiety disorder symptoms measured with the Social Phobia Inventory (SPIN). Scores go from 0 (no social anxiety symptoms) to 68 (severe social anxiety symptoms).
Panic disorder symptoms | Panic Disorder Severity Scale - Self Report version (PDSS-SR) will be administered after 8 weeks of treatment.
  Improvement of panic disorder symptoms measured with the Panic Disorder Severity Scale - Self Report version (PDSS-SR). Scores go from 0 (no panic symptoms) to 4 (severe panic symptoms).
Functioning | Sheehan Disability Scale (SDS) will be administered after 8 weeks of treatment.
  Improvement of functioning measured with the Sheehan Disability Scale (SDS). Scores go from 0 (no functional impairment) to 10 (severe functional impairment).
Sustained response | Clinical Global Impression - Improvement scale (CGI-I) will be administered two weeks after the end of the treatment.
  Treatment response will be defined as a score of 1 or 2 on the Clinical Global Impression - Improvement scale (CGI-I).
  CGI-I scores range from 0 to 7. Zero corresponds to "not assessed". Low scores correspond to improvement, high scores correspond to worsening.
Sustained remission | Clinical Global Impression - Severity scale (CGI-S) will be administered two weeks after the end of the treatment.
  Remission will be defined as a score of 1 or 2 on the Clinical Global Impression - Severity scale (CGI-S).
  CGI-S scores range from 0 to 7. Zero corresponds to "not assessed". Low scores correspond to mild and high scores correspond to severe.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Freire, MD PhD, Principal Investigator — Department of Psychiatry, Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No